CLINICAL TRIAL: NCT03359096
Title: Cardiovascular Endpoints for Obstructive Sleep Apnea With Twelfth Nerve Stimulation (CARDIOSA-12): A Randomized, Sham-Controlled, Double-Blind, Crossover Trial
Brief Title: Hypoglossal Nerve Stimulation on Cardiovascular Outcomes
Acronym: CARDIOSA-12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: American Heart Association (Other); American Academy of Sleep Medicine (Other)
Responsible Party: Principal Investigator, Raj Dedhia, MD, Associate Professor of Otorhinolaryngology: Head and Neck Surgery, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 834158
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Results first posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep apnea; Tongue stimulation; Cardiovascular function
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Washout Period 1 (Study Week 1): The patient will not use Hypoglossal Nerve Stimulation (HGNS) for 1 week. Randomization Visit (Study Week 2): The patient will be randomized to sub-therapeutic HGNS (sham) or therapeutic HGNS (treatment) for 28 days. Sympathetic and Vascular testing (Study Week 6). Washout Period 2 (Study Week 6-7): The patient will not use HGNS for 7 days. The patient will be switched to the other intervention arm (treatment to sham vs. sham to treatment) for 28 days. Sympathetic and Vascular testing (Study Week 11).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Therapeutic HGNS (Experimental): Therapeutic Hypoglossal Nerve Stimulation (HGNS). Prior to enrollment in this study, the HGNS will have been implanted as part of clinical care, and a therapeutic voltage setting will have been determined via overnight sleep study.
  Interventions: Device: Therapeutic HGNS
- Subtherapeutic 'Sham' HGNS (Sham Comparator): Sham threshold determination will be performed as follows. The patient will be in a reclined position with the mouth open while nasal breathing. Stimulation will be increased from 0.1V up by 0.1V until bulk tongue motion is detected without obvious protrusion. This process is repeated twice and the average value is used to determine "sham-HGNS". The electrode configuration will remain consistent between the patient's therapeutic and sham thresholds.
  Interventions: Device: Subtherapeutic 'Sham' HGNS

INTERVENTIONS:
Device: Therapeutic HGNS — Prior to enrollment in this study, the HGNS will have been implanted as part of clinical care, and a therapeutic voltage setting will have been determined via overnight sleep study The pulse generator, using technology from cardiac pacemakers, utilizes the signal from the pressure sensor for timing of stimulation to the tongue nerve. Patient will undergo activation of the implanted device one month post-operatively. A functional threshold (in volts) is obtained based on tongue motion during device stimulation. For the next month, the patient will have steadily increased stimulation strength by 0.1V every 2-3 nights within the preset range until the upper limit is reached.
  Other Names: Hypoglossal Nerve Stimulation
  Arms: Therapeutic HGNS
Device: Subtherapeutic 'Sham' HGNS — Sham threshold determination will be performed as follows. The patient will be in a reclined position with the mouth open while nasal breathing. Stimulation will be increased from 0.1V up by 0.1V until bulk tongue motion is detected without obvious protrusion. This process is repeated twice and the average value is used to determine "sham-HGNS". The electrode configuration will remain consistent between the patient's therapeutic and sham thresholds
  Other Names: Sham Hypoglossal Nerve Stimulation
  Arms: Subtherapeutic 'Sham' HGNS

SUMMARY:
A new, well-tolerated treatment for obstructive sleep apnea - tongue stimulation - is a device which opens the airway during sleep and can provide treatment for patients unable to use the mask and hose treatment. The study will evaluate the effect of this new treatment on blood pressure and heart-related measures to see if it lowers patients' risk of heart problems.

DETAILED DESCRIPTION:
Obstructive sleep apnea, repetitive airway blockage during sleep, affects 1 in 10 Americans. If left untreated, it results in decreased quality of life and increased risk of heart problems. Only half of these people are able to use the main treatment, continuous positive airway pressure (CPAP) therapy, which involves wearing a mask and hose at night. A new, well-tolerated treatment - tongue stimulation - is a device which opens the airway during sleep and can provide treatment for patients unable to use the mask and hose treatment. The study will evaluate the effect of this new treatment on blood pressure and heart-related measures to see if it lowers patients' risk of heart problems.

ELIGIBILITY:
All patients recruited into the study will have already been implanted with the Inspire® HGNS device.

Additional Inclusion Criteria include:

* As tolerating the therapeutic level during sleep can take time (weeks to months), all patients must be able to use the device at the therapeutic setting (> 20 hours/week for > 1 month) prior to enrollment, based on compliance data.
* All patients will be English-speaking and able to give written informed consent.

Exclusion Criteria include:

* Inspire® remote Model 2500 or later is required. Patients with older remotes are not candidates due to limited adherence monitoring capabilities.
* Patients who have fallen asleep while driving resulting in accident or "near miss" accident within 1 year prior to HGNS implantation.
* Actively using positive airway pressure (PAP) therapy for treatment of OSA.
* Patients in whom the difference between sham and therapeutic voltages is less than 30% the therapeutic voltage.
* Pregnant women will be excluded.*

  * Women of childbearing potential must NOT be pregnant or plan on becoming pregnant. This study involves temporarily stopping treatment of obstructive sleep apnea, which may harm the fetus. If applicable, the patient will need to take a urine pregnancy test after enrollment (prior to washout #1), and again prior to washout #2.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj C Dedhia, MD, MSCR, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Dedhia RC, Quyyumi AA, Park J, Shah AJ, Strollo PJ, Bliwise DL. Cardiovascular endpoints for obstructive sleep apnea with twelfth cranial nerve stimulation (CARDIOSA-12): Rationale and methods. Laryngoscope. 2018 Nov;128(11):2635-2643. doi: 10.1002/lary.27284. Epub 2018 Sep 8. PMID 30194765
- [Derived] Dedhia RC, Bliwise DL, Quyyumi AA, Thaler ER, Boon MS, Huntley CT, Seay EG, Tangutur A, Strollo PJ, Gurel N, Keenan BT. Hypoglossal Nerve Stimulation and Cardiovascular Outcomes for Patients With Obstructive Sleep Apnea: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2024 Jan 1;150(1):39-48. doi: 10.1001/jamaoto.2023.3756. PMID 38032624

RESULTS

PARTICIPANT FLOW:
Groups:
- Therapeutic HGNS, Then Subtherapeutic 'Sham' HGNS: Therapeutic Hypoglossal Nerve Stimulation (HGNS): Prior to enrollment in this study, the HGNS will have been implanted as part of clinical care, and a therapeutic voltage setting will have been determined via overnight sleep study The pulse generator, using technology from cardiac pacemakers, utilizes the signal from the pressure sensor for timing of stimulation to the tongue nerve. Patient will undergo activation of the implanted device one month post-operatively. A functional threshold (in volts) is obtained based on tongue motion during device stimulation. For the next month, the patient will have steadily increased stimulation strength by 0.1V every 2-3 nights within the preset range until the upper limit is reached.
  Subtherapeutic 'Sham' HGNS: Sham threshold determination will be performed as follows. The patient will be in a reclined position with the mouth open while nasal breathing. Stimulation will be increased from 0.1V up by 0.1V until bulk tongue motion is detected without obvious protrusion. This process is repeated twice, and the average value is used to determine "sham-HGNS". The electrode configuration will remain consistent between the patient's therapeutic and sham thresholds.
- Subtherapeutic 'Sham' HGNS, Then Therapeutic HGNS: Subtherapeutic 'Sham' HGNS: Sham threshold determination will be performed as follows. The patient will be in a reclined position with the mouth open while nasal breathing. Stimulation will be increased from 0.1V up by 0.1V until bulk tongue motion is detected without obvious protrusion. This process is repeated twice and the average value is used to determine "sham-HGNS". The electrode configuration will remain consistent between the patient's therapeutic and sham thresholds.
  Therapeutic HGNS: Prior to enrollment in this study, the HGNS will have been implanted as part of clinical care, and a therapeutic voltage setting will have been determined via overnight sleep study The pulse generator, using technology from cardiac pacemakers, utilizes the signal from the pressure sensor for timing of stimulation to the tongue nerve. Patient will undergo activation of the implanted device one month post-operatively. A functional threshold (in volts) is obtained based on tongue motion during device stimulation. For the next month, the patient will have steadily increased stimulation strength by 0.1V every 2-3 nights within the preset range until the upper limit is reached.
Period: HGNS Washout (1 Week)
Arm/Group | Therapeutic HGNS, Then Subtherapeutic 'Sham' HGNS | Subtherapeutic 'Sham' HGNS, Then Therapeutic HGNS
Started | 31 | 32
Completed | 31 | 31
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: First Intervention (4 Weeks)
Arm/Group | Therapeutic HGNS, Then Subtherapeutic 'Sham' HGNS | Subtherapeutic 'Sham' HGNS, Then Therapeutic HGNS
Started | 31 | 31
Completed | 29 | 31
Not Completed | 2 | 0
Not completed — Death | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: HGNS Washout (1 Week)
Arm/Group | Therapeutic HGNS, Then Subtherapeutic 'Sham' HGNS | Subtherapeutic 'Sham' HGNS, Then Therapeutic HGNS
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Therapeutic HGNS, Then Subtherapeutic 'Sham' HGNS | Subtherapeutic 'Sham' HGNS, Then Therapeutic HGNS
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Therapeutic HGNS, Then Subtherapeutic 'Sham' HGNS: Therapeutic Hypoglossal Nerve Stimulation (HGNS): Prior to enrollment in this study, the HGNS will have been implanted as part of clinical care, and a therapeutic voltage setting will have been determined via overnight sleep study The pulse generator, using technology from cardiac pacemakers, utilizes the signal from the pressure sensor for timing of stimulation to the tongue nerve. Patient will undergo activation of the implanted device one month post-operatively. A functional threshold (in volts) is obtained based on tongue motion during device stimulation. For the next month, the patient will have steadily increased stimulation strength by 0.1V every 2-3 nights within the preset range until the upper limit is reached.
  Subtherapeutic 'Sham' HGNS: Sham threshold determination will be performed as follows. The patient will be in a reclined position with the mouth open while nasal breathing. Stimulation will be increased from 0.1V up by 0.1V until bulk tongue motion is detected without obvious protrusion. This process is repeated twice, and the average value is used to determine "sham-HGNS". The electrode configuration will remain consistent between the patient's therapeutic and sham thresholds.
  *The trial's total enrollment was 63 patients; however, 3 patients were consented & enrolled but did not complete the entirety of study procedures. One patient was consented and enrolled but withdrew prior to intervention assignment, and two patients withdrew prior to crossover.
- Subtherapeutic 'Sham' HGNS, Therapeutic HGNS: Subtherapeutic 'Sham' HGNS: Sham threshold determination will be performed as follows. The patient will be in a reclined position with the mouth open while nasal breathing. Stimulation will be increased from 0.1V up by 0.1V until bulk tongue motion is detected without obvious protrusion. This process is repeated twice and the average value is used to determine "sham-HGNS". The electrode configuration will remain consistent between the patient's therapeutic and sham thresholds.
  Therapeutic HGNS: Prior to enrollment in this study, the HGNS will have been implanted as part of clinical care, and a therapeutic voltage setting will have been determined via overnight sleep study The pulse generator, using technology from cardiac pacemakers, utilizes the signal from the pressure sensor for timing of stimulation to the tongue nerve. Patient will undergo activation of the implanted device one month post-operatively. A functional threshold (in volts) is obtained based on tongue motion during device stimulation. For the next month, the patient will have steadily increased stimulation strength by 0.1V every 2-3 nights within the preset range until the upper limit is reached.
  *The trial's total enrollment was 63 patients; however, 3 patients were consented & enrolled but did not complete the entirety of study procedures. One patient was consented and enrolled but withdrew prior to intervention assignment, and two patients withdrew prior to crossover.
- Total: Total of all reporting groups
Arm/Group | Therapeutic HGNS, Then Subtherapeutic 'Sham' HGNS | Subtherapeutic 'Sham' HGNS, Therapeutic HGNS | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (7.5) | 67.1 (11.8) | 67.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 18 | 20 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26 | 29 | 55
  Black | 3 | 0 | 3
  Hispanic | 0 | 1 | 1
  Asian | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.6 (4.9) | 27.9 (4.2) | 28.7 (4.6)
Pre-Implant Apnea-Hypopnea Index (AHI) [Mean (Standard Deviation); unit: events/hour] | 34.4 (15.0) | 31.9 (14.9) | 33.1 (14.9)

OUTCOME MEASURES:

1. Primary Outcome: Mean 24-Hour Systolic Ambulatory Blood Pressure Values
Description: Patients will undergo 24-hour ambulatory blood pressure testing (ABP) using a noninvasive, portable device. The monitor is programmed to record blood pressure every 30 minutes. The patient will be asked to record bedtime and wake time to corroborate the sleep and wake time from the recorder. Mean 24-hour systolic ambulatory blood pressure values will be calculated.
Time Frame: Study Week 6, Day 1; study Week 11, Day 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Therapeutic HGNS | Subtherapeutic 'Sham' HGNS
Number analyzed (Participants) | 60 | 60
mmHg | 122.8 (11.8) | 123.0 (10.8)

2. Secondary Outcome: Mean 24-Hour Diastolic Ambulatory Blood Pressure Values
Description: Patients will undergo 24-hour ambulatory blood pressure testing (ABP) using a noninvasive, portable device. The monitor is programmed to record blood pressure every 30 minutes. The patient will be asked to record bedtime and wake time to corroborate the sleep and wake time from the recorder. Mean 24-hour diastolic ambulatory blood pressure values will be calculated.
Time Frame: Study Week 6, Day 1; study Week 11, Day 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Therapeutic HGNS | Subtherapeutic 'Sham' HGNS
Number analyzed (Participants) | 60 | 60
mmHg | 71.9 (7.8) | 72.1 (7.0)

3. Secondary Outcome: Mean Nocturnal Systolic and Diastolic Ambulatory Blood Pressure Values
Description: Patients will undergo ambulatory blood pressure testing (ABP) using a noninvasive, portable device. The patient will be asked to record bedtime and wake time to corroborate the sleep and wake time from the recorder. Mean sleep systolic and diastolic ambulatory blood pressure values will be calculated.
Time Frame: Study Week 6, Day 1; study Week 11, Day 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Therapeutic HGNS | Subtherapeutic 'Sham' HGNS
Number analyzed (Participants) | 60 | 60
mmHg
  SLEEP systolic blood pressure | 115.0 (14.6) | 114.8 (14.0)
  SLEEP diastolic blood pressure | 65.8 (9.1) | 66.3 (8.7)

4. Secondary Outcome: Mean Muscle Sympathetic Nerve Activity (MSNA) Frequency (Bursts/Minute)
Description: The peroneal nerve will be located with transcutaneous stimulation and a tungsten microelectrode will be inserted into the nerve, and a reference electrode will be inserted 1-2 cm from the recording electrode. Nerve signals will be preamplified, amplified, filtered, rectified, and integrated to obtain a mean voltage display of sympathetic nerve activity that is recorded. Muscle sympathetic bursts will be identified by visual inspection and expressed as burst frequency (bursts per minute).
  MSNA was only performed on 7 patients at Emory University, prior to the trial being transferred to the University of Pennsylvania. This is due to there being no research collaborators available at the University of Pennsylvania to capture MSNA as part of this trial. There is insufficient data gathered to make meaningful claims regarding this outcome measure.
Time Frame: Study Week 6, Day 2; Study Week 11, Day 2
Population: MSNA was only performed on 7 patients at Emory University, prior to the trial being transferred to the University of Pennsylvania. For MSNA performed during Therapeutic HGNS arm, 3 patients did not have analyzable MSNA data. For MSNA performed during subtherapeutic 'Sham' HGNS arm, 2 patients did not have analyzable MSNA data.
Measure: Mean (Standard Deviation); unit: bursts/minute
Arm/Group | Therapeutic HGNS | Subtherapeutic 'Sham' HGNS
Number analyzed (Participants) | 4 | 5
bursts/minute | 20.2 (10.6) | 17.6 (5.8)

5. Secondary Outcome: Mean Muscle Sympathetic Nerve Activity (MSNA) Tonal Activity (Units/Minute)
Description: The peroneal nerve will be located with transcutaneous stimulation and a tungsten microelectrode will be inserted into the nerve, and a reference electrode will be inserted 1-2 cm from the recording electrode. Nerve signals will be preamplified, amplified, filtered, rectified, and integrated to obtain tonal activity (units/minute).
  MSNA was only performed on 7 patients at Emory University, prior to the trial being transferred to the University of Pennsylvania. This is due to there being no research collaborators available at the University of Pennsylvania to capture MSNA as part of this trial. There is insufficient data gathered to make meaningful claims regarding this outcome measure.
Time Frame: Study Week 6, Day 2; Study Week 11, Day 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units/minute
Arm/Group | Therapeutic HGNS | Subtherapeutic 'Sham' HGNS
Number analyzed (Participants) | 4 | 5
units/minute | 29.6 (15.1) | 7.0 (23.9)

6. Secondary Outcome: Mean Pre-Ejection Period (PEP)
Description: A patient will be fitted with Impedance Cardiography (ICG) Noninvasive Cardiac Output Module that will record the ECG (Electrocardiogram) and the ICG (Impedance cardiography) continuously during a 10-minute period. PEP will be calculated as the average interval (milliseconds) from the onset of left ventricular depolarization, reflected by the Q-wave onset in the ECG to the opening of the aortic valve, reflected by the B-point in the ICG signal. A significant difference in PEP to be a 10 millisecond increase from baseline.
Time Frame: Study Week 6, Day 2; Study Week 11, Day 2
Population: Due to COVID-19 related resource constraints and/or poor signal quality acquisition, several PEP measurements were not included for analysis.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Therapeutic HGNS | Subtherapeutic 'Sham' HGNS
Number analyzed (Participants) | 51 | 50
milliseconds | 105.7 (16.5) | 105.4 (16.8)

7. Secondary Outcome: Mean Flow-mediated Dilation (FMD)
Description: The brachial artery of the nondominant arm will be imaged using a high-resolution ultrasound transducer. A blood pressure cuff on the forearm will be inflated to suprasystolic pressures to produce 5 min of ischemia. On cuff deflation, imaging will be performed to measure FMD. Brachial artery FMD will be calculated as (post-ischemia diameter - baseline diameter) / (baseline diameter) x 100.
Time Frame: Study Week 6, Day 2; Study Week 11, Day 2
Population: Due to COVID-19 related resource constraints and/or poor signal quality acquisition, several FMD measurements were not included for analysis.
Measure: Mean (Standard Deviation); unit: % of dilation from baseline
Arm/Group | Therapeutic HGNS | Subtherapeutic 'Sham' HGNS
Number analyzed (Participants) | 43 | 42
% of dilation from baseline | 6.65 (4.38) | 6.79 (5.03)

8. Secondary Outcome: Mean Peripheral Arterial Stiffness (PAS)
Description: Following a rest period of 10 minutes with subjects in a supine position in a quiet, temperature-controlled room, blood pressure will be measured 3 times at 5-minute intervals by an automatic device. The standard metric of peripheral arterial stiffness (PAS) is carotid-femoral pulse wave velocity (PWV), which will be estimated using the Sphygmocor device® (Atcor Medical, Sydney, Australia).
  PAS was only captured on 21 patients at Emory University and the University of Pennsylvania. This is due to our cardiovascular research collaborators at the University of Pennsylvania indicating they would no longer be able to support our research study due to their own COVID-19 related resource constraints. There is insufficient data gathered to make meaningful claims regarding this outcome measure.
  PAS is reported as changes in pulse wave velocity, with a meters/second unit measure.
Time Frame: Study Week 6, Day 2; Study Week 11, Day 2
Population: For PAS performed during Therapeutic HGNS arm, 2 patients did not have analyzable PAS data.
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Therapeutic HGNS | Subtherapeutic 'Sham' HGNS
Number analyzed (Participants) | 19 | 21
meters/second | 11.1 (6.2) | 9.8 (2.8)

9. Secondary Outcome: Mean Psychomotor Vigilance Test (PVT) Reciprocal Reaction Time
Description: Patients will perform the neurobehavioral test on a specially calibrated (for timing precision) and designated laptop in a quiet room in the outpatient setting. Each patient will perform a unique version of the psychomotor vigilance test to assess psychomotor speed.
  The trial's protocol was amended to begin capturing neurobehavioral measures like the PVT at the University of Pennsylvania, as part of a new collaboration with research collaborators in the Department of Psychiatry. PVT is a validated instrument to capture attention, and response time on this cognitive test is reported as reciprocal milliseconds or 1/milliseconds.
Time Frame: Study Week 6, Day 2; Study Week 11, Day 2
Population: PVT was only captured on 43 patients following the trial's transfer from Emory University to the University of Pennsylvania. This was due to a new collaboration between the Department of Otorhinolaryngology & the Department of Psychiatry to investigate changes in cognitive status for obstructive sleep apnea patients being treated with HGNS.
Measure: Mean (Standard Deviation); unit: 1/milliseconds
Arm/Group | Therapeutic HGNS | Subtherapeutic 'Sham' HGNS
Number analyzed (Participants) | 43 | 43
1/milliseconds | 4.01 (0.47) | 3.97 (0.51)

10. Secondary Outcome: Mean Digit Symbol Substitution Test (DSST) Reaction Time
Description: Patients will perform the neurobehavioral test on a specially calibrated (for timing precision) and designated laptop in a quiet room in the outpatient setting. Each patient will perform a unique version of the digit symbol substitution test to assess processing speed.
  The trial's protocol was amended to begin capturing neurobehavioral measures like the DSST at the University of Pennsylvania, as part of a new collaboration with research collaborators in the Department of Psychiatry. DSST is a validated instrument to capture visual tracking and working memory, and response time on this cognitive test is reported in milliseconds.
Time Frame: Study Week 6, Day 2; Study Week 11, Day 2
Population: DSST was only captured on 43 patients following the trial's transfer from Emory University to the University of Pennsylvania. This was due to a new collaboration between the Department of Otorhinolaryngology & the Department of Psychiatry to investigate changes in cognitive status for obstructive sleep apnea patients being treated with HGNS.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Therapeutic HGNS | Subtherapeutic 'Sham' HGNS
Number analyzed (Participants) | 43 | 43
milliseconds | 1846.64 (355.5) | 1893.57 (428.1)

ADVERSE EVENTS:
Time Frame: through study completion, an average duration of 10 weeks.
Groups:
- Therapeutic HGNS; Subtherapeutic 'Sham' HGNS: Therapeutic Hypoglossal Nerve Stimulation (HGNS): Prior to enrollment in this study, the HGNS will have been implanted as part of clinical care, and a therapeutic voltage setting will have been determined via overnight sleep study The pulse generator, using technology from cardiac pacemakers, utilizes the signal from the pressure sensor for timing of stimulation to the tongue nerve. Patient will undergo activation of the implanted device one month post-operatively. A functional threshold (in volts) is obtained based on tongue motion during device stimulation. For the next month, the patient will have steadily increased stimulation strength by 0.1V every 2-3 nights within the preset range until the upper limit is reached.
  Subtherapeutic 'Sham' HGNS: Sham threshold determination will be performed as follows. The patient will be in a reclined position with the mouth open while nasal breathing. Stimulation will be increased from 0.1V up by 0.1V until bulk tongue motion is detected without obvious protrusion. This process is repeated twice, and the average value is used to determine "sham-HGNS". The electrode configuration will remain consistent between the patient's therapeutic and sham thresholds.
  *The trial's total enrollment was 63 patients; however, 3 patients were consented & enrolled but did not complete the entirety of study procedures. One patient was consented and enrolled but withdrew prior to intervention assignment, and two patients withdrew prior to crossover.
Arm/Group | Therapeutic HGNS | Subtherapeutic 'Sham' HGNS
All-Cause Mortality (participants affected / at risk) | 0/60 | 1/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

LIMITATIONS AND CAVEATS:
* partially therapeutic effect of sham HGNS
* recruitment of patients with dramatic symptomatic improvement with HGNS was challenging as these patients declined to be without treatment for 6 out of 10 weeks
* HGNS is appropriate for a select subset of OSA patients, limiting generalizability of study findings.
* baseline AHI was obtained from patient medical records, other baseline outcome measurements (ABPM, PEP, FMD) were not obtained
* excluded severely excessively sleepy OSA patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT03359096/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT03359096/ICF_001.pdf